CLINICAL TRIAL: NCT05354999
Title: Effects of Different Combinations of Performance-enhancing Supplements on High Intensity Exercise Performance
Brief Title: Effects of Combinations of Performance-enhancing Supplements on Exercise Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Morten Hostrup, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: COCKTAIL
Record Dates: First submitted 2022-04-18; First posted 2022-05-02 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Exercise; Performance; Supplementation
MeSH Terms: conditions — Motor Activity | interventions — Sodium Bicarbonate; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine (Experimental): Subjects ingest creatine monohydrate daily.
  Interventions: Dietary Supplement: Sodium bicarbonate and caffeine
- Placebo (Placebo Comparator): Subjects ingest placebo daily.
  Interventions: Dietary Supplement: Sodium bicarbonate and caffeine

INTERVENTIONS:
Dietary Supplement: Sodium bicarbonate and caffeine — On experimental days subjects ingest a combination of sodium bicarbonate, caffeine and placebo.

SUMMARY:
The purpose of the study is to investigate the effect of combinations of creatine monohydrate, sodium bicarbonate and caffeine on exercise performance and fatigability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* VO2max of >50 ml/min/kg for men and >45 ml/min/kg for women
* Performs endurance training >3 times per week

Exclusion Criteria:

* Chronic disease deemed by the study responsible medical doctor to interfere with any part of the study
* Smoking
* Chronic use of prescription medicine deemed by the study responsible medical doctor to interfere with any part of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Work performed (kJ/Watt) | Measured at each trial throughout the study, on average 4 weeks
  Work performed during a 6 minute time trial

SECONDARY OUTCOMES:
Work performed (kJ/Watt) | Measured at each trial throughout the study, on average 4 weeks
  Work performed during a 15 second sprint test
Muscle strength (Nm) | Measured at each trial throughout the study, on average 4 weeks
  Maximal voluntary isometric contraction of m. quadriceps femoris

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided